CLINICAL TRIAL: NCT04076696
Title: Clinical Evaluation of Primary Sampling Scatter Correction for Chest Tomosynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC1822; 18-1144 (Other: UNC IRB); 1R21CA216780-01A1 (NIH)
Record Dates: First submitted 2019-08-27; First posted 2019-09-03 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple
Keywords: Chest; Lung; Tomography; Scatter
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Scatter corrected s-DCT (Experimental): The study scan, s-DCT and correction scan, will be performed within two weeks of the patient's clinical evaluations by chest CT and x-ray. The study scan may be done within 2 weeks prior or two weeks following standard of care imaging. There cannot be any intervening therapies or procedures (i.e. biopsy or excision of lesions) done in between the standard of care (SOC) imaging and the s-DCT. All patients will have a breath held s-DCT scan in an anterior-posterior direction.
  Interventions: Device: Scatter corrected s-DCT

INTERVENTIONS:
Device: Scatter corrected s-DCT — All patients will have a breath held s-DCT scan in an anterior-posterior direction

SUMMARY:
This is a study that will evaluate the utility of a scatter reduction technique in reducing dose and increasing the sensitivity of stationary digital chest tomosynthesis (s-DCT) in the detection of lung lesions.

DETAILED DESCRIPTION:
Digital tomosynthesis is an imaging modality that produces 3D sectional information using x-ray projections acquired over a limited scanning angle. Scatter is known to be the primary source of image degradation in x-ray based imaging.

The investigators have developed an approach that measures scatter through a low dose (3% of the conventional scan) scatter measurement technique. Preliminary studies have shown that scatter reduction in DCT can significantly improve quality. The approach will characterize the reader confidence in lung nodule detection in a scatter corrected chest tomosynthesis imaging approach as compared to the conventional chest tomosynthesis.

Fifty (50) patients who have undergone a clinical non-contrast CT with lung nodules will be asked to have an s-DCT (scan) within 4 weeks (+/- 2 week) of their clinical CT with no intervening procedures or therapies (i.e. biopsy of lung nodules). Investigators will then perform a reader study to evaluate the radiologist reader confidence in images generated from the scatter reduction technique versus more conventional chest tomosynthesis imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known lung lesion(s)
* Patients having undergone a chest CT
* Patients 18 years of age and older
* Patients able to provide informed consent

Exclusion Criteria:

* Patients who may not fit on a 35 x 35 detector (BMI > 35)
* Planned procedures or therapies during study (in between SOC scans and study scan on s-DCT) (biopsy or removal of lung lesion)
* Any woman who is pregnant, has reason to believe she is pregnant, or is lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2021-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ertan Pamuklar, MD, Principal Investigator — UNC Hospitals
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Scatter Corrected s-DCT
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Scatter Corrected s-DCT
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 32
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Reader Confidence in s-DCT Images Compared to Conventional CT (Units on a Scale)
Description: Readers will rate their confidence in images from the experimental modality (sDCT with scatter correction) as compared to the conventional scan (chest CT with x-ray) on a 7 point Likert scale (-3 to 3) based on ability to identify lesion(s) present comparing each modality. A value of -3 is significantly less confident in the s-DCT representation 0 is the same confidence in modalities, and 3 is significantly more confident in the s-DCT representation compared to the conventional. Each individual will have a single value per reader. Two readers compared each scan. The overall reader preference between modalities was calculated by determining the mean value.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Scatter Corrected s-DCT
Number analyzed (Participants) | 38
Units on a scale | -0.43 (0.62)

2. Secondary Outcome: Sensitivity of s-DCT Images (Percentage of Positive Scans)
Description: Sensitivity will be defined as the ability of s-DCT images to detect lesions positively identified on gold standard CT images.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of positive scans
Arm/Group | Scatter Corrected s-DCT
Number analyzed (Participants) | 38
percentage of positive scans | 0.407 [0.224 to 0.612]

ADVERSE EVENTS:
Time Frame: Adverse events occurring during the participants' participation in the study visit were collected directly following imaging for 30 minutes post imaging.
Arm/Group | Scatter Corrected s-DCT
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-12): https://cdn.clinicaltrials.gov/large-docs/96/NCT04076696/Prot_SAP_000.pdf